CLINICAL TRIAL: NCT06611670
Title: Outcomes of High Vs Physiological Intraocular Pressure During Cataract Surgery Using ACTIVE SENTRY
Acronym: ACTIVESENTRY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Samir Jabbour, Ophthalmologist, Assistant clinical professor, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-11959
Record Dates: First submitted 2024-09-22; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Cataract; Cataract Surgery; Cataract Bilateral
Keywords: Active Sentry; cataract surgery; cataracts; High intra-ocular pressure; central corneal thickness; intraocular pressure; phacoemulsification; safety profile; physiological IOP
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Interventional single-masked pair-eye design clinical trial, single-center, single-surgeon. Eyes will be block-randomized as to which surgery they will receive first (high vs low IOP phacoemulsification). 76 eyes of 38 patients will be included in this study. For each patient, one eye will be randomized to receive phacoemulsification with high IOP (Group 1), and the other eye will receive phacoemulsification with physiological IOP (Group 2). This way, each patient will receive both treatments, one for each eye, which will allow us to do paired analyses.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cataract surgery with Active Sentry (Experimental): Cataract surgery with low IOP values (32mmHg)
  Interventions: Device: Cataract surgery with Active Sentry
- High IOP (Active Comparator): Cataract surgery with high IOP (60mmHg) which is the average pressure at which cataract surgery is being performed currently
  Interventions: Procedure: Traditional cataract surgery

INTERVENTIONS:
Device: Cataract surgery with Active Sentry — Surgical instrument that detects changes in intraocular pressure and allows rapid feedback to stabilize pressure during cataract surgery.
  Arms: Cataract surgery with Active Sentry
Procedure: Traditional cataract surgery — Cataract surgery performed with high intraocular pressures
  Arms: High IOP

SUMMARY:
Cataract surgery is a widely performed procedure across the world that helps restore vision in many patients suffering from cataracts. Irrigation is an essential component of the surgery. Fluid is constantly circulated to help regulate temperature as heat is generated with ultrasound energy, to minimize tissue trauma, and to create an intraocular pressure (IOP) sufficient to keep the anterior chamber (AC) stable. In parallel, aspiration brings the components of the cataract closer to the surgical instrument. A balance between irrigation and aspiration during surgery is essential to maintain stability in the AC. However, an ideal flow rate, which influences IOP during surgery, is yet to be determined. Most recent studies with Centurion Active Sentry show that there is similar efficiency between higher and lower IOP settings. Traditionally, high-flow rates have been used in advanced cataracts and are believed to make space in the AC. However, they are known to create fluid turbulence and are associated with risks of tissue damage, including cell loss in one of the cornea's layers. High IOP during surgery has also been shown to cause damage to the optic nerve as well as to the retina. Distorting and stretching the AC during phacoemulsification have also been associated with increased pain experienced by the patient. Comfort can be achieved by lowering pressure levels. Low-flow rates have a better safety profile, reduce IOP and pressure fluctuations while offering equal efficiency, including comparable surgical time. Using central corneal thickness (CCT) as an indicator of corneal trauma, it has been shown that patients that have had surgery with low-flow rates present no change in the CCT postoperatively as opposed to patients in the high-flow rates. As less fluid turbulence is created with low-flow rates, there is decreased risk of fragment contact with the cornea's inner surface, thus reducing cell loss. Alcon Laboratories, Inc. developed Active Fluidics which allows to stabilize intraocular pressure and prevent IOP fluctuations as well as IOP surges during surgery. It is now further equipped with the Active Sentry handpiece which is integrated to the surgical instrument and acts as a sensor to pressure variation. It allows rapid feedback to maintain a stable AC. Our research project aims to assess the outcomes following phacoemulsification done with physiological IOP with the help of the Active Sentry handpiece compared to traditional high IOP levels.

DETAILED DESCRIPTION:
Cataract surgery is a widely performed procedure across the world that helps restore vision in many patients suffering from cataracts. The surgery has known many improvements across time and continues to do so. Irrigation is an essential component of the surgery. Fluid is constantly being circulated to help regulate temperature as heat is generated with the use of ultrasound energy, to minimize tissue trauma, and to create an intraocular pressure sufficient to keep the anterior chamber stable. In parallel, aspiration brings the components of the cataract closer to the surgical instrument. A balance between irrigation and aspiration during surgery is essential to maintain stability in the anterior chamber. However, an ideal flow rate, which influences intraocular pressure (IOP) during surgery, is yet to be determined. Most recent studies with Centurion Active Sentry (maintaining vacuum and aspiration rates the same) show that there is similar efficiency between higher and lower IOP settings. Traditionally, high-flow rates have been used in advanced cataracts and are believed to increase the space in the anterior chamber. However, they are known to create fluid turbulence and are associated with risks of tissue damage, including cell loss in the endothelial layer of the cornea. High intra-ocular pressure during surgery has also been shown to cause damage to the optic nerve as well as to the retina. Distorting and stretching the anterior chamber during phacoemulsification have also been associated with increased pain experienced by the patient. Comfort can be achieved by lowering pressure levels. Low-flow rates have a better safety profile, reduce IOP and pressure fluctuations while offering equal efficiency, including comparable surgical time. Using central corneal thickness (CCT) as an indicator of corneal trauma, it has been shown that patients that have had surgery with low-flow rates present no change in the CCT postoperatively while patients in the high-flow rates show signs of corneal damage as well as greater anterior segment inflammation. As less fluid turbulence is created with low-flow rates, there is decreased risk of fragment contact with the cornea's inner surface, thus reducing cell loss. Alcon Laboratories, Inc. developed Active Fluidics which allows to stabilize intraocular pressure and prevent IOP fluctuations as well as IOP surges during surgery. It is now further equipped with the Active Sentry handpiece which is integrated to the surgical instrument and acts as a sensor to pressure variation. It allows rapid feedback to maintain a stable anterior chamber. Our research project aims to assess the outcomes following phacoemulsification done with physiological IOP with the help of the Active Sentry handpiece compared to traditional high IOP levels.

ELIGIBILITY:
Inclusion Criteria:

* No prior ocular surgery including corneal refractive surgery
* Bilateral visually significant cataract, similar in density (LOCS III grade 2+), undergoing uncomplicated cataract surgery
* Equal dilated pupil size ≥6mm, no use of pupil expansion devices
* Axial length 22-26mm, refractive error between -5.00D to +5.00D and cylinder ≤ 3.00D, normal K values <47.00D
* Axial eye length cannot vary by more than 0.4 mm between eyes of an individual patient
* Normal CCT range 540µm ± 50

Exclusion Criteria:

* History of corneal disease or dystrophies
* Media opacification for reasons other than cataract
* Compromised zonular integrity or stability.
* Retinal and retinal vascular pathologies, age-related macular degeneration
* Glaucoma
* Patients with uncontrolled systematic diseases, including hypertension, diabetes, systemic cardiovascular diseases, and hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Central corneal thickness at 1 day postoperatively | 1 day postoperatively
  Using central corneal thickness (CCT) as an indicator of corneal trauma, it has been shown that patients that have had surgery with low-flow rates present no change in the CCT postoperatively. CCT will be measured using a pachymetry (Normal CCT range 540µm ± 50).

SECONDARY OUTCOMES:
Volume of balanced salt solution used during surgery | During surgery
  Volume of balanced salt solution as measured by the Active Sentry Centurion machine
Total ultrasound time and total aspiration time | During surgery
  Total ultrasound time and total aspiration time as measured by the Active Sentry Centurion machine
Endothelial cell loss (inner surface of the cornea) | At month 1 and month 3 postoperatively.
  Endothelial cell count measured by specular microscopy
Central corneal thickness | 1 week, 1 month and 3 months postoperatively
  Using central corneal thickness (CCT) as an indicator of corneal trauma, it has been shown that patients that have had surgery with low-flow rates present no change in the CCT postoperatively. CCT will be measured using a pachymetry (Normal CCT range 540µm ± 50).
Corneal clarity | Day 1, week 1, month 1 and month 3 postoperatively
  Measured uring the Pentacam corneal densitometry

OTHER OUTCOMES:
Visual acuity | Day 1, week 1, month 1, and month 3 postoperatively
  Evaluated using a Snellen chart
Low contrast evaluation | Day 1, week 1, month 1, and month 3 postoperatively
  Evaluated using the CSV-1000 Contrast Sensitivity chart with glare
Intraocular pressure | Day 1, week 1, month 1, and month 3 postoperatively
  Measured using the Goldmann Applanation Tonometer
Cystoid macular edema | 1 month postoperatively
  Evaluated using the Macular Optical Coherence Tomography (OCT)
Rate of reverse pupillary block | 1 day, 1 week, 1 month and 3 months postoperatively
  Evaluated using slit lamp examination
Posterior capsular tear | During surgery
  Complication during cataract surgery
Posterior capsular rupture | During surgery
  Complication during cataract surgery

CONTACTS AND LOCATIONS:
Overall Officials: Samir Jabbour, MD,CM,FRCSC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao Y, Li X, Tao A, Wang J, Lu F. Intraocular pressure and calculated diastolic ocular perfusion pressure during three simulated steps of phacoemulsification in vivo. Invest Ophthalmol Vis Sci. 2009 Jun;50(6):2927-31. doi: 10.1167/iovs.08-2996. Epub 2009 Jan 24. PMID 19168897
- [Background] Vasavada AR, Praveen MR, Vasavada VA, Vasavada VA, Raj SM, Asnani PK, Garg VS. Impact of high and low aspiration parameters on postoperative outcomes of phacoemulsification: randomized clinical trial. J Cataract Refract Surg. 2010 Apr;36(4):588-93. doi: 10.1016/j.jcrs.2009.11.009. PMID 20362850